CLINICAL TRIAL: NCT07297797
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of HRS-9563 in Patients With Mild to Moderate Hypertension
Brief Title: Phase II Clinical Study of HRS-9563 in Patients With Mild to Moderate Hypertension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9563-201
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Mild to Moderate Hypertension
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: HRS-9563 or Placebo Injection; low dose (Experimental)
  Interventions: Drug: HRS-9563 Injection; Drug: sodium chloride injection
- Treatment group B: HRS-9563 or Placebo Injection; Intermediate dose (Experimental)
  Interventions: Drug: HRS-9563 Injection; Drug: sodium chloride injection
- Treatment group C: HRS-9563 or Placebo Injection; Medium to high dose (Experimental)
  Interventions: Drug: HRS-9563 Injection; Drug: sodium chloride injection
- Treatment group D: HRS-9563 or Placebo Injection; high dose (Experimental)
  Interventions: Drug: HRS-9563 Injection; Drug: sodium chloride injection

INTERVENTIONS:
Drug: HRS-9563 Injection — HRS-9563 Injection
Drug: sodium chloride injection — sodium chloride injection

SUMMARY:
This study aims to evaluate the efficacy and safety of HRS-9563 in patients with mild to moderate hypertension, and to explore its appropriate dosage.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily signs the informed consent form.
2. Male or female, aged ≥ 18 years and ≤ 75 years;
3. Patients with mild to moderate hypertension;
4. At the Screening and Baseline periods, the mean sitting office systolic blood pressure is > 130 mmHg, and the 24-hour mean systolic blood pressure assessed by ABPM at Screening is ≥ 130 mmHg and < 160 mmHg.

Exclusion Criteria:

1. Secondary hypertension;
2. Orthostatic hypotension;
3. Type 1 diabetes or poorly controlled type 2 diabetes;
4. Occurrence of any cardiovascular or cerebrovascular event within 6 months prior to screening;
5. Presence of uncontrolled severe arrhythmia within 6 months prior to screening;
6. Suspected allergy to the investigational drug or any of its components;
7. Other diseases requiring Renin-Angiotensin-Aldosterone System (RAAS) inhibitor therapy, besides hypertension;
8. Any blood biochemical indicator during screening or baseline did not meet the standards in the exclusion criteria;
9. Use of any medication affecting blood pressure within 4 weeks prior to screening, or planned use during the study period;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour mean systolic blood pressure assessed by ABPM at month 6 | at 6 months after initiation of administration

SECONDARY OUTCOMES:
Change from baseline in 24-hour mean systolic blood pressure assessed by ABPM at month 3 | at 3 months after initiation of administration
Change from baseline in 24-hour mean systolic blood pressure assessed by ABPM at month 9 | at 9 months after initiation of administration
Change from baseline in 24-hour mean diastolic blood pressure assessed by ABPM at month 3 | at 3 months after initiation of administration
Change from baseline in 24-hour mean diastolic blood pressure assessed by ABPM at month 6 | at 6 months after initiation of administration
Change from baseline in 24-hour mean diastolic blood pressure assessed by ABPM at month 9 | at 9 months after initiation of administration
Change from baseline in mean sitting office systolic blood pressure at month 3; | at 3 months after initiation of administration
Change from baseline in mean sitting office systolic blood pressure at month 6; | at 6 months after initiation of administration
Change from baseline in mean sitting office systolic blood pressure at month 9; | at 9 months after initiation of administration
Change from baseline in mean sitting office diastolic blood pressure at month 3; | at 3 months after initiation of administration
Change from baseline in mean sitting office diastolic blood pressure at month 6; | at 6 months after initiation of administration
Change from baseline in mean sitting office diastolic blood pressure at month 9; | at 9 months after initiation of administration

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided